CLINICAL TRIAL: NCT04211025
Title: Screening for Poverty and Related Social Determinants and Intervening to Improve Knowledge of and Links to Resources (SPARK) Pilot Study
Brief Title: Screening for Poverty and Related Social Determinants to Improve Knowledge of and Links to Resources (SPARK) Pilot Study
Acronym: SPARK Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Project ID 1532
Record Dates: First submitted 2019-05-28; First posted 2019-12-26 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2019-12

CONDITIONS: Primary Care
Keywords: Sociodemographic Screening; Income; Primary Care; Social Needs

STUDY DESIGN:
Intervention Model Description: Intervention
  Our intervention consists of two parts:
  1. Routine screening for sociodemographics and social needs such as poverty
  2. Intervening when poverty is identified through linkage to a trained staff member who uses a Benefits Screening Tool to identify benefits that the patient is entitled to, and then provides support
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modest (Experimental): This approach is feasible to integrate into workflows of a wide-range of clinics, and should have a minimal impact on human resources. Materials and strategies to support staff in this work will be provided. .
  Interventions: Other: Modest
- Intensive (Experimental): This approach is more robust, and requires a greater commitment of human resources.
  Interventions: Other: Intensive

INTERVENTIONS:
Other: Modest — The modest intervention consists of a 30-minute appointment (by phone or in-person) with the designated staff using the Benefits Screening Tool , and a plan is developed. At 4 weeks, the designated staff follows-up with a phone call or email.
  Arms: Modest
Other: Intensive — The intensive intervention consists of a 30-minute appointment with the designated staff using the Benefits Screening Tool , and a plan is developed. At 4 weeks, a follow-up appointment is booked for 30 minutes, and progress on the plan is assessed. At 12 weeks after the initial meeting, the designated staff follows-up with a phone call or email.
  Arms: Intensive

SUMMARY:
Research question and objectives This pilot study will help us answer the following research question: Is it feasible to conduct a large cluster randomized controlled trial (RCT) of an intervention that consists of routine screening for poverty and related social determinants and intervening in Canadian primary care clinics, and what is the sample size required?

Our objectives include:

1. to collect data on the feasibility of recruiting clinics for a large cluster randomized controlled trial (RCT)
2. to collect data on the acceptability and feasibility of integrating a standardized socio-demographic data collection tool, including screening for poverty, within diverse primary care clinic workflows
3. collect data on the acceptability and feasibility of "modest" and "intensive" interventions on poverty (discussed below)
4. collect data on the recruitment rate of patients, to assist with calculating the sample size for a larger cluster RCT
5. collect data on the intervention effect size of the "modest" and "intensive" interventions on income and health outcomes to assist with calculating the sample size for a larger cluster RCT .

DETAILED DESCRIPTION:
Rationale Research carried out by members of the study team has found that routine socio-demographic data collection in primary care has significant potential. Such data could be used to better tailor care to a patient's social context, improve diagnostic accuracy by incorporating social determinants as risk factors, identify inequities in the uptake of health services and in health outcomes, stimulate the development of new programs, and advance research. However, a standard set of questions has not yet been developed in Canada. Significant challenges remain to implementation of routine socio-demographic data collection, particularly around patient engagement, staff training, and support to make use of data collected, including adjustment for non-response bias. Existing work has also found that health providers and organizations lack evidence-based interventions to address social needs, particularly poverty. Work to date by the study team has found that a prototype financial benefit tool could be integrated into clinic workflow, particularly if the right staff person was administering it and following up with patients, and approximately 17% of patients had received a financial benefit after 1 month. No study to date has examined the longer-term impact of such a tool on income and health. It is not known whether a "modest" intervention, with the tool integrated into a clinic visit and brief follow-up, would be as effective as a more "intensive" intervention, with a dedicated visit to use the tool and multiple follow-up visits

ELIGIBILITY:
Inclusion Criteria:

Patients: The inclusion criteria are as follows:

1. A patient who completed the sociodemographic and social needs survey in their primary care organization.
2. Answers "Yes" to the question "Do you have difficulty making ends meet at the end of the month?" and answers "Yes" to the question "Our clinic is part of a study of how to help patients who may be eligible for financial benefits. Would you like to take part?"
3. Able to provide consent
4. Age is greater than or equal to 18
5. Able to converse in English
6. Able to be reached via telephone, email, or through coordination with their clinic site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Access to Additional Benefits | 2 months follow-up
  The primary outcome measure will be whether or not participants accessed additional benefits and/or increased income as a result of participating in the study. This will be determined through the phone surveys with participants, conducted by the study team
Access to Additional Benefits | 4 months follow-up
  The primary outcome measure will be whether or not participants accessed additional benefits and/or increased income as a result of participating in the study. This will be determined through the phone surveys with participants, conducted by the study team

SECONDARY OUTCOMES:
Implementation data (sociodemographic and social needs survey) | Through study completion, up to 1 year
  Number of people completing the sociodemographic and social needs survey
Implementation data (income screening question) | Through study completion, up to 1 year
  Number of people who answer positively to the income screening question
Implementation data (income assistance indication) | Through study completion, up to 1 year
  Number of people who answer indicate they would like assistance with income
Implementation data (recruitment and staff time) | Through study completion, up to 1 year
  Number of people recruited to the study; time required for staff to complete the Benefit Screening Tool and follow-up
Implementation data (staff time) | Through study completion, up to 1 year
  Time required for staff to complete the Benefit Screening Tool and follow-up
Patient self-reported stress as part of qualitative interview | 2 months follow-up
  Stress Levels (Never, Rarely, Sometimes, Often, Always)
Patient self-reported quality of life on the PROMIS Global 10 Generic Health Questionnaire | 2 months follow-up
  Quality of Life (Excellent, Very Good, Good, Fair, Poor)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pinto, MD MSc, Principal Investigator — Unity Health Toronto
Locations (6):
- Canada (6):
  - Queen's Family Health Team, Kingston, Ontario
  - Platinum Medical Clinic, Scarborough Village, Ontario
  - New Family Medicine Network, North York Family Health Team, Toronto, Ontario
  - Southeast Toronto Family Health Team, Toronto, Ontario
  - East End Community Health Centre, Toronto, Ontario
  - Access Alliance, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No